ID: Pro00103863

Identifying the Optimal Neural Target for Misophonia Interventions

NCT04348591

Approved Study econsent FINAL reference date 2.4.2022



# **CONCISE SUMMARY**

We are doing this study to learn more about the difference between misophonia and general problems reducing emotional arousal.

People in this study will have 1-2 screening visit(s) that includes obtaining medical and psychiatric interviews, questionnaires about function and emotions, and a task where you will listen and rate how you feel after listening to several different sounds.

Next we will ask participants to return for an MRI scan, where we will look at what happens in their brains while they are listening to potentially distressing sounds.

Everyone who joins this study will learn how to use *Regulation Strategies* (learning to think differently about emotional situations) and then practice them during exposure to potentially distressing sounds while receiving different types of *neurostimulation*. Neurostimulation involves placement of a wire coil shaped like an 8 on the scalp that produces very small electric currents in the part of the brain that is closest to the coil.

Participation in the study may take up to 2 months and includes 3-4 visits.

About 2 out of 1000 people may have a seizure during the neurostimulation. The most common side effect is headache.

If you are interested in learning more about this study, please continue to read below.

The purpose of this e-consent form is to give you the information you will need to help you decide whether or not to be in the study.

We are asking you to take part in this research study because you have expressed interest in participating in our Misophonia studies or have difficulties managing your emotions. You may ask any questions about the purpose of the research, what we would ask you to do, the possible risks and benefits, your rights as a volunteer, and anything else about the research or this form that is not clear. When all of your questions have been answered, you can decide if you want to be in the study or not. This process is called 'informed consent'. You will receive a copy of this signed and dated e-consent form for your records.

Research studies are voluntary and include only people who choose to take part. Please read this consent form carefully and take your time making your decision. As the study staff discusses this consent form with you, please ask him/her to explain any words or information that you do not clearly understand. We encourage you to talk with your family and friends before you decide to take part in this research study. The nature of the study, risks, inconveniences, discomforts, and other important information about the study are listed below.



Please tell the study staff if you are taking part in another research study.

**Dr.** Andrada D. Neacsiu will conduct the study that is paid for by a grant from the Misophonia Research Fund (MRF) awarded by the REAM foundation. Portions of *Dr. Neacsiu's* salary is covered by MRF.

# WHO WILL BE MY DOCTOR ON THIS STUDY?

If you decide to participate, Doctors Andrada Neacsiu and Noreen Bukhari-Parlakturk will be your doctors for the study and will be in contact with your regular health care provider if needed during the study or after.

# WHY IS THIS STUDY BEING DONE?

Misophonia, the inability to tolerate certain repetitive distressing sounds that are common, is gaining recognition as an impairing condition. It is not a well-understood condition and there are no known treatments. In this study we examine what separates misophonia from other types of emotional distress. We plan to examine changes in brain activity during presentation and regulation of misophonic versus distressing sounds. We plan to alter activity in key areas of the misophonia brain circuitry with the goal to identify new misophonia interventions.

The type of neuromodulation used in the study is repetitive transcranial magnetic stimulation (rTMS), a procedure which involves placement of an electromagnetic coil over the scalp that produces very small electric currents in the part of the brain that is closest to the coil. rTMS is a noninvasive and painless treatment that is approved by the Food and Drug Administration (FDA) for the treatment for depression only. In this study, we will use rTMS differently than what has been approved for by the FDA but within safety guidelines.

Using rTMS in studies for conditions other than depression is investigational. The word "investigational" means the study device is still being tested in research studies and is not approved by the U.S. Food and Drug Administration (FDA) for this condition.

# HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

About 60 people will take part in this study at Duke. Thirty adults who report significant misophonic distress and 30 who report high emotional dysregulation. We may enroll up to 200 people in order to have 60 people complete the study.

**DUHS IRB** IRB NUMBER: Pro00103863

IRB REFERENCE DATE: 02/04/2022 IRB EXPIRATION DATE: 02/26/2023



# WHAT IS INVOLVED IN THE STUDY?

| | Assessment Day(s) | MRI Day | Neurostimulation<br>Day |
|---|---|---|---|
| Consent discussion | <b>A</b> | | - |
| Medical and treatment history | <b>A</b> | | <b>A</b> |
| Questionnaires | <b>A</b> | <b>A</b> | <b>A</b> |
| Computer tasks with physiological recording | <b>A</b> | <b>A</b> | <b>A</b> |
| Interview | <b>A</b> | | |
| Urine test (females of childbearing potential) | | <b>A</b> | <b>A</b> |
| Regulation Strategies Training | | <b>A</b> | <b>A</b> |
| rTMS | | | <b>A</b> |
| Brain imaging | | <b>A</b> | |

These activities are described in detail below.

# Assessment Appointment (1-2 Visits):

If you choose to take part in this study, you will first be asked to sign and date this e-consent form. You have already completed the telephone or online screening, but we are not yet sure if you will be eligible for the study. Today's visit will last between 1 and 4 hours.

During your first study visit (today) you will talk with an assessor about your medical and mental health history. Questions will include your drug use, psychological problems, how you cope with stress, ways in which you tend to think about yourself, and how you get along with others.

We will ask you about your treatment history, including any medications you may be currently taking (for example, prescription medications, over-the-counter medications and vitamins).

During this visit, we will also ask you to complete a number of questionnaires that tell us about your difficulties managing emotions, misophonia, COVID impact, general mental health and distress, functional impairment, anxiety, depression, and coping.

We would like you to keep any other treatment that you are part of consistent throughout the study. If you are enrolled in psychotherapy, you cannot change or stop the therapy during the study. Also, you can be on medication for mental health problems as long as there have been no changes in your medication in the past month and you agree not to make any changes in medication throughout the study (with the exception of a medical emergency).

If you have recently participated in other studies here in our clinic, you may not have to answer all of the interview questions that we normally ask during this visit. Instead, we will use the answers that you gave in your other recent visit when we review the data for this study. The



study staff will review the results of the visit to decide if you continue to qualify for the study.

If you do not qualify to stay in the study, your time and your participation will be complete at this point.

If you do qualify, you will next be scheduled to complete a sound task at a separate in person visit. During the in person sound task appointment, you will be asked to rate your distress level to a sample of sounds including sounds from the International Affective Digitized Sound System. We will record your facial expressions when you hear these sounds and will monitor your skin conductance (i.e., how sweaty your fingers get) while you are listening to the sounds. The facial recording is optional. Please note, it will not be done during visits that occur when COVID safety guidelines are being followed. You may complete this in person task without the facial recording. You will need to complete the sound task before your imaging appointment.

Please indicate below if you are willing to allow researchers to record your facial expressions during the in person sound task.

I am willing to allow the researchers to video-record my face during the in-person sound task.

I am NOT willing to allow the researchers to video-record my face during the sound task OR I am not willing to attend the sound task in person.

If you do qualify, we will then schedule you for the next appointment. Sometimes the interviews and questionnaires can last longer than expected. If this first visit is lasting longer than planned, we may have to finish it on a second day. If that is the case, you will finish the interviews or the self-report scales before the next session. We will only ask you to finish the visit and questionnaires on the second day if you qualify for the study.

We will video record or audio record you as part of this study to make sure the research staff are doing the study procedures correctly. If you are not willing to be video-or audio-recorded, please indicate so below (you will still be eligible to be in the study).

Recordings will be kept strictly confidential and will be directly recorded on Duke office computers/laptops using a web camera directly connected to the computer's hard drive. The recordings will then be immediately transferred from the computer's/laptop's hard drive to the Duke protected hard drive that is maintained and secured by Duke in the Department of Psychiatry and Behavioral Sciences. The folder that will contain these video/audio recordings is protected and only members of the study team who are listed as key study personnel can access them. The video/audio-recordings may be reviewed by the key research and clinical staff members in Dr. Neacsiu's team, and may also be used for training within Dr. Neacsiu's lab of new research staff, if you agree. At the end of the study, you may review the recordings and



delete any portions you don't want us to save. You have the right to come in and erase any parts of the recording, but you do not have a right to copy our recordings or any of our research material. These recordings will be destroyed at least six years after the study is completed.

Please indicate below whether or not you are willing to be audio or video-recorded as part of this research study.

I am willing to allow the researchers to video-record the interviews to see if the experimenter is following the protocol correctly.

I am willing to allow the researchers to ONLY audio-record the interviews to see if the experimenter is following the protocol correctly.

I am NOT willing to allow the researchers to record the interviews.

# **MRI Session:**

As soon as possible after the 1-2 assessment visit(s), we will have the neuroimaging session (MRI Day) which will last about 2-3 hours. We will meet in the lobby of the main Duke hospital and walk together to MRI facility (4-minute walk). If you are a female of childbearing potential, we will ask you to provide a urine sample to check if you are pregnant. We will not continue with the MRI visit if the pregnancy test is positive for your own safety. The Magnetic Resonance Imaging (MRI) instrument being used in this study has a part that is not commercially available and is considered investigational and is being used for research purposes only.

We will train you in the Regulation Strategies (i.e., ways to think about the sounds that help you feel less distressed). We will practice on several sounds that are not your own distressing sounds.

We will also ask you to complete some online questionnaires.

If you have never had a brain MRI, you will have the option to have a "mock scan" to familiarize you with the sights and sounds of the procedure using a practice MRI machine.

During the MRI portion of the session, you will lie on your back upon a narrow bed that will be pushed into the MRI machine. The MRI technician will provide padding for your head and knees to make you more comfortable while lying down.

If you are uncomfortable or feel pain because of lying down, please tell the technician right away. The technician will also place a respiration belt on your chest, two electrodes on your fingers, and a clip on another finger so we can monitor your skin conductance, breathing and pulse during the scan. The technician will position your head inside a head tube, and the platform will be pushed inside the MRI machine. You will be able to communicate with the technician during the MRI using a microphone and speaker in the MRI machine.



While you are in the scanner you will be presented with a series of sounds and asked to rate your level of distress. This portion of the study will take about 1.5 hours.

# **Neurostimulation Session:**

When you return to the lab for the neurostimulation session, we will meet in a different building. This session will last 3-4 hours. If you are a female of childbearing potential, we will ask you to provide a urine sample to check if you are pregnant. We do this to ensure your safety.

Before you come in, we will check whether the brain neurostimulation we are planning is safe for you. The study team may review your medical history and some of the forms you completed during the assessment day. Based on the study team's review and the urine pregnancy test we will decide whether it is safe for you to continue with the study.

The use of rTMS in this study is considered investigational.

We will ask you about any changes in your medications, drug, caffeine, alcohol, & nicotine use on that day, your sleep habits, and current pain, physical distress, and drowsiness levels. You will also be retrained in the Regulation Strategies.

Establishing dose of brain stimulation and rTMS protocol. The rTMS equipment includes an electric stimulator and a wire coil. Turning the stimulator on and off produces brief electrical currents in the coil, and these currents create a magnetic field around that coil. The wire coil is shaped like an '8', coated in plastic, and is a little larger than a piece of notebook paper. When the coil is held close to the head, it generates a magnetic field which can induce very small electric currents in the part of the brain that is closest to the coil. These currents are similar to the currents that the neurons (brain cells) in the brain create when communicating with each other.

Before applying rTMS, the study doctors will need to decide what "dose" of stimulation to use for you by establishing your personal "motor threshold." To establish this threshold, we will first place the stimulator over the part of your brain that controls the motor activity in your left or right hand. You will hear a clicking sound and feel a tapping sensation at your scalp. The stimulator will be adjusted to give just enough energy so that the motor region of the brain sends signals to your hand muscles, to make your hand twitch. The lowest amount of energy required to make your hand twitch is called the "motor threshold." Everyone has a different motor threshold. This will take about 15 minutes.

Using your brain imaging data, we will identify several areas for brain stimulation. The rTMS stimulation will be applied over one of these pre-determined areas of your brain. We will also connect you to our physiological recording equipment and record your skin conductance and heart rate baseline for five minutes. Once this set up is complete, the experimental task will begin. You will be instructed to engage in different methods of thinking differently to either regulate or feel emotions associated with negative and neutral sounds while receiving different



types of neurostimulation. You will be able to take a break in between each portion of the task. Before each break, we will ask you to rate your emotional distress and level of dissociation during the previous task. At the end of the session, we will ask you to complete an online questionnaire about your experience in the study, your current level of distress, emotions, and any side effects that you might have from neurostimulation. The neurostimulation session will last 3-4 hours.

# HOW LONG WILL I BE IN THIS STUDY?

Your participation in the study may last up to 2 months. This includes 3-4 visits: the screening visit(s), the MRI session, and the neurostimulation session.

We will try to have all procedures completed within two weeks but may extend to 8 weeks if finding times for you to come in is difficult.

# WHAT ARE THE RISKS OF THE STUDY?

As a result of being in this study, you are at risk for the following side effects. You should discuss these with the study doctor and your regular health care provider if you choose.

# **Risks of rTMS:**

The most serious known risk of TMS is seizures. TMS procedures come with a very low risk of seizures. Out of over 10,000 people given various forms of TMS to date, 16 people (less than 0.2%) have had a seizure. TMS can produce a seizure when a series of pulses is given at high power and when repeated series of pulses are given extremely close together.

This study will use only levels of TMS that are within safety guidelines. Levels of TMS that fall within the safety guidelines have not been associated with seizures in people who have been evaluated medically and undergone the motor threshold test. No seizures have occurred in normal volunteers with the dosage of TMS used in this study.

To minimize this risk, we will medically screen you for any of medical reasons that could lead to seizures. For example, persons with epilepsy cannot be in this study. You will be watched carefully during the TMS for any signs of seizure or muscle twitching. In spite of these precautions, there is a chance that you will experience a seizure.

Should this occur, emergency facilities are available. If you have a seizure, you may require hospital admission and follow-up neurological evaluation. Having had a seizure may make it difficult for you to obtain medical insurance, future employment, and to drive. It is not known whether having had one seizure will make a person more prone to have future seizures. Should you have a seizure caused by TMS in this protocol, we will provide you with a letter stating the seizure was caused by a research procedure.

The most commonly reported side effect of TMS a "muscle-tension" type headache. About three

DUHS IRB

IRB NUMBER: Pro00103863

7



out of ten people may experience a headache with the types of TMS used in this study. We will make every effort to reduce any discomfort.

If a headache occurs, it usually starts during or immediately after the TMS and lasts from minutes to hours. The headache usually goes away with standard over-the-counter pain medications. You may also have neck pain. You may also experience some discomfort on your head where the coil is placed. This is due to contraction of scalp muscles. If you experience pain and discomfort, we may apply lidocaine or a thin plastic sheet to help with the uncomfortable sensation.

Numbness of the face lasting for a short time has also been reported in rare instances and may last for several weeks after receiving the procedure. Fainting is considered a rare side effect of TMS and has been reported in people who faint during blood draws. If you experience fainting, you will be withdrawn from the study and have your blood pressure monitored until it returns to a healthy level.

The clicking noises produced by the TMS procedure are loud enough to be damaging to your ears. You will therefore be required to wear earphones and listen to white noise during the TMS procedures.

Additional rare side effects of TMS are dizziness, memory problems, trouble concentrating, and acute mood changes. If these happen, they usually do not last long and will resolve without need for treatment.

There may be other risks that are currently unknown. The long-term effects of rTMS are not known.

# Risks of regulation strategies and behavioral assessment:

It is possible that you may experience some unpleasant thoughts or emotions from the interviews, questionnaires and/or tasks on the computer. However, we have no reason to believe that any unpleasant thoughts or emotions will last long after the experiment is over. Some of the questions we will ask you as part of this study may make you feel temporarily uncomfortable, as they have to do with psychological problems such as depression, or anxiety.

You may refuse to answer any of the questions and you may take a break at any time during the study. If you are feeling very upset during an assessment interview or the sound task, a trained staff member will be available to talk with you about these feelings.

If at any time during the interviews or the procedures you have strong thoughts of suicide, you should notify the study staff and a trained professional will be available to talk. The trained study staff will work with you to address these suicidal thoughts and if you are at imminent risk of



suicide after the conversation, you will be taken to the nearest hospital emergency room (for example: Duke ER).

There is also a potential risk of loss of confidentiality. Every effort will be made by the study staff to keep your information confidential; however, this cannot be guaranteed.

If you have any medical adverse events (a bad effect) after leaving the TMS laboratory, please contact the Duke operator at 919-684-8111 and have Dr. Noreen Bukhari-Parlakturk paged. If you have any psychological adverse events, please have Dr. Andrada Neacsiu paged at the same number.

# Risks of MRI Scan:

Magnetic resonance imaging (MRI) uses a magnet and radio waves to make diagnostic medical images of the body. There have been no ill effects reported from exposure to the magnetism or radio waves used in this test. However, it is possible that harmful effects could be recognized in the future. A known risk is that the magnet could attract certain kinds of metal. Therefore, we will carefully ask you about metal within your body, including medical implants, devices such as pacemakers and internal defibrillators, or certain dyes found in tattoos. We will also keep the examining room locked so that no one carrying metal objects can enter while you are in the scanner.

If there is any question about potentially hazardous metal within your body, you will not undergo the MRI. This may exclude you from participation in this research study. The MRI involves entering a large room in which a magnet is present. You will be placed on a narrow bed and then slid into a small tunnel approximately 6 feet in length and 25 inches in diameter. You will be asked to lie still for about one hour on this bed. You will hear a loud machine-like noise. You may be asked to have a harmless monitoring device applied during the MRI. During the MRI, you can have voice contact and physical contact with someone in attendance if you desire. Let the study doctor know if you have a fear of enclosed spaces.

# **Reproductive Risks:**

**For women of who can get pregnant:** The effects of the MRI and TMS on a developing pregnancy are not known. In addition, the changes that women who are pregnant or breastfeeding undergo can affect the responses to some of the tests. Women who are pregnant or who are planning a pregnancy are not allowed to participate in the study.

If you are a woman who can get pregnant, a urine pregnancy test will be done on the day of the MRI scan and the rTMS session, and it must be negative before you can continue in this study.

Although there are no potential risks to a developing pregnancy in between the MRI or TMS sessions, if you become pregnant between sessions you will not be able to continue in the study. Therefore, we recommend that you either abstain completely from vaginal intercourse until your

DUHS IRB

IRB NUMBER: Pro00103863

IRB REFERENCE DATE: 02/04/2022 IRB EXPIRATION DATE: 02/26/2023



last session, or use an effective method of contraception for the same length of time. Effective methods include partner vasectomy, bilateral tubal ligation, intrauterine devices (IUDs), hormonal methods, or barrier methods (condoms, diaphragms, cervical caps) with spermicide.

# ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

This study may be of no direct benefit to you, but you will help improve our knowledge about misophonia and emotional dysregulation. A possible benefit is that the study could help develop personalized strategies for you to use to feel better when upset, but this cannot be guaranteed. We hope that in the future the information learned from this study will benefit other people with your condition.

# WHAT IF WE LEARN ABOUT NEW FINDINGS OR INFORMATION DURING THE

You will be given any new information gained during the course of the study that might affect your willingness to continue. If any unexpected abnormalities are found that might pose a significant health risk to you, Dr. Neacsiu will inform you so that you may seek follow up medical consultation with a doctor of your choosing.

# POSSIBLE DISCOVERY OF FINDINGS RELATED TO MEDICAL IMAGING

It is possible that the MRI component of this study will identify information about you that was previously unknown, such as disease status or risk. This research scan is not a medical diagnostic test.

There are no plans to provide this information to you or your physician unless there is an unexpected finding on the scan that indicates a possible need for follow-up testing. This is rare, occurring in only about 3 of every 1000 people scanned. If this happens, your scan will be reviewed by a physician or the MRI technician, who may recommend further diagnostic testing. If this happens, the physician or MRI technician will discuss this with you and you will be asked for separate permission for the follow-up and further testing outside of this research study. The possible costs associated with this follow-up and/or further testing will be discussed with you at that time.

# WHAT ALTERNATIVES ARE THERE TO PARTICIPATION IN THIS STUDY?

You do not have to participate in this study to get treatment for your mental health problems. Currently available treatments include many types of psychotherapy and medications. Please talk to your doctor about these and perhaps other options.

# WILL MY INFORMATION BE KEPT CONFIDENTIAL?

Participation in research involves some loss of privacy. We will do our best to make sure that information about you is kept confidential, but we cannot guarantee total confidentiality. Your personal

**DUHS IRB** 

IRB NUMBER: Pro00103863

IRB REFERENCE DATE: 02/04/2022 IRB EXPIRATION DATE: 02/26/2023



information may be viewed by individuals involved in this research and may be seen by people including those collaborating, funding, and regulating the study. We will share only the minimum necessary information in order to conduct the research. Your personal information may also be given out if required by law. Except when required by law, you will not be identified by name, social security number, address, telephone number, or any other direct personal identifier in study records disclosed outside of Duke University Health System (DUHS).

All paper data and research forms will be kept in a secure locked cabinet in Dr. Neacsiu's office and will only be made available to members of the research team for this study. Your name and other personal identifying information will not be stored in the computer system databases that store your ratings, and thus individuals who might gain unauthorized access to your ratings will not know your identity.

Video recordings which could contain identifiable information will be destroyed no more than 6 years after the study is completed.

Your name and other personal identifying information will not be used in any scientific reports of this study, and will not be made available to representatives from award groups. Some people or groups who receive your health information might not have to follow the same privacy rules.

Once your information is shared outside of DUHS, we cannot guarantee that it will remain private. If you decide to share private information with anyone not involved in the study, the federal law designed to protect your health information privacy may no longer apply to the information you have shared. Other laws may or may not protect sharing of private health information.

Your records may be reviewed in order to meet federal or state regulations. Reviewers may include the representatives from the sponsor, and the Duke University Health System Institutional Review Board. If either of these groups review your research record, they may also need to review your entire medical record (if you receive your medical care at DUHS).

The study results will be retained in your research record for at least six years after the study is completed. At that time, either the research information not already in your medical record will be destroyed or information identifying you will be removed from such study results at DUHS. Any research information in your medical record will be kept indefinitely.

The study results will be combined with results from other subjects and given to the FDA to support applications to use rTMS. All reasonable efforts will be made to keep your identity confidential. Because of the need to release safety information to third parties, absolute confidentiality cannot be guaranteed. This information may be further disclosed by the sponsors of this study Duke University and MRF. If disclosed by the sponsor, the information is no longer covered by federal privacy regulations.



Another risk to your confidentiality comes from someone intercepting emails we send to you. We will keep the information in e-mails brief, but an e-mail breach would get your e-mail address connected to a Duke study. No other information should be apparent if there is a breach. The link to the online survey is generic and does not "remember" your previous answers. Therefore, if someone else accesses the link from your e-mail they will not be able to see any answers that you have entered. We will use REDCAP, a Duke approved platform, to collect your information

A description of this clinical trial will be available on <a href="www.ClinicalTrials.gov">www.ClinicalTrials.gov</a>, as required by US law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

# WHAT ARE THE COSTS?

There will be no additional costs to you as a result of being in this study.

#### WHAT ABOUT COMPENSATION?

You will be compensated up to \$250 for your participation and will be given a parking pass or a bus pass to cover your travel to Duke during days when you have in person visits. All payments will be made at the end of your participation.

When you finish the assessment day, and you are not eligible to participate in the full study, you will receive \$20 plus a parking pass at the Duke Hospital parking garage or a bus pass (up to \$3) to cover the

cost of parking or bus fare, if applicable. If you are eligible, you will receive \$40 for completing the interview and questionnaire portion. For completing the sound task in person with physiological data collection, you will receive \$35 plus a parking or bus pass, if applicable. Thus, you will receive a total of \$75 for the initial 1-2 assessment visit(s).

After the initial screening day, compensation for the study depends upon the procedures that you complete. You will get \$75 for completing the imaging session. You will be paid \$10 if you attempt to complete the MRI session but do not complete it (because of detected pregnancy or claustrophobia). You will also be compensated for parking at this visit.

If TMS is medically appropriate, you will be paid \$100 for the neurostimulation day plus parking or bus pass. If you cannot tolerate the TMS procedure and stop early, you will be compensated \$20 plus a parking pass or bus pass.

For eligible participants, all payments will be done at the end of the study.



# WHAT ABOUT RESEARCH RELATED INJURIES?

Immediate necessary medical care is available at Duke University Medical Center in the event that you are injured as a result of your participation in this research study. However, there is no commitment by Duke University, Duke University Health System, Inc., or your Duke physicians to provide monetary compensation or free medical care to you in the event of a study-related injury.

For questions about the study or research-related injury, contact Dr. Neacsiu at 919-684-6714 during regular business hours. If outside regular business hours, please contact the Duke operator at 919-684-8111 and have Dr. Andrada Neacsiu paged.

# WHAT ABOUT MY RIGHTS TO DECLINE PARTICIPATION OR WITHDRAW FROM THE STUDY?

You may choose not to be in the study, or, if you agree to be in the study, you may withdraw from the study at any time. If you withdraw from the study, no new data about you will be collected for study purposes unless the data concern an adverse event (a bad effect) related to the study. If such an adverse event occurs, we may need to review your entire medical record. All data that have already been collected for study purposes, and any new information about an adverse event related to the study, will be sent to the study sponsor.

Your decision not to participate or to withdraw from the study will not involve any penalty or loss of benefits to which you are entitled, and will not affect your access to health care at Duke. However, if you decide to stop participating, we encourage you to talk to a staff member so we can best assist you to find additional services if needed.

Nonparticipation or withdrawal from this study will not affect your job status if you are a Duke employee and will not affect your grades if you are a Duke student. If you do decide to withdraw, we ask that you contact Dr. Neacsiu in writing and let her know that you are withdrawing from the study. Her mailing address is Box 3026, Duke University Medical Center, Durham, NC 27710 or you can email her at <a href="mailto:Andrada.neacsiu@duke.edu">Andrada.neacsiu@duke.edu</a>.

We will tell you about new information that may affect your health, welfare, or willingness to stay in this study. Your doctor may decide to take you off this study if your condition gets worse, if you have serious side effects, or if the study team determines that it is no longer in your best interest to continue

# WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or a research-related injury, or if you have problems, concerns, questions

or suggestions about the research, contact Dr. Andrada Neacsiu at 919-684-6714 during regular business hours, or the Duke operator outside of business hours at 919-684-8111 to have Dr. Neacsiu paged.

DUHS IRB

IRB NUMBER: Pro00103863



For questions about your rights as a research participant, or to discuss problems, concerns or suggestions related to the research, or to obtain information or offer input about the research, contact the Duke University Health System Institutional Review Board (IRB) Office at (919) 668-5111.

# STATEMENT OF CONSENT

"The purpose of this study, procedures to be followed, risks and benefits have been explained to me. I have been allowed to ask questions, and my questions have been answered to my satisfaction. I have been told whom to contact if I have questions, to discuss problems, concerns, or suggestions related to the research, or to obtain information or offer input about the research. I have read this consent form and agree to be in this study, with the understanding that I may withdraw at any time. I have been told that I will be given a signed and dated copy of this consent form."

| 0 | "Yes, I have read the | e consent document | and I wish to | narticipate in | the study " |
|---|---|---|---|---|---|
| | 1 cb, 1 mayo roud un | consent document | una i wish to | participate in | me staay. |

<sup>&</sup>quot;Yes, I have read the consent document and I DO NOT wish to participate in the study."